CLINICAL TRIAL: NCT06129526
Title: Study of the Effect of Eicosapentaenoic Acid (EPA) on Markers of Atherothrombosis in Patients With Type-2 Diabetes
Brief Title: Study of the Efficacy and Safety of EPA in Patients With Type-2 Diabetes
Acronym: SEASIDE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ioannina (Other)
Collaborators: LIBYTEC Pharmaceutical S.A. (Unknown)
Responsible Party: Principal Investigator, Alexandros Tselepis, Emeritus Professor of Clinical Biochemistry, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EPA-UOI 2023
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Type 2; Hypertriglyceridemia; Diabetes Mellitus
Keywords: Atherothrombosis; Biomarkers; Coronary Artery Disease (CAD); Corn oil; Eicosapentaenoic acid; Endothelial cells; Inflammation; Omega-3; Platelets; Polyunsaturated Fatty Acids (PUFAs)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertriglyceridemia; Diabetes Mellitus; Thrombosis; Coronary Artery Disease; Inflammation | interventions — Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EPAVasc 2g (Active Comparator)
  Interventions: Dietary Supplement: EPAVasc
- EPAVasc 2g x 2 (Active Comparator)
  Interventions: Dietary Supplement: EPAVasc
- Corn Oil (Placebo Comparator)
  Interventions: Dietary Supplement: Corn Oil

INTERVENTIONS:
Dietary Supplement: EPAVasc — EPAVasc: 1,875mg EPA / 125mg DHA / 3.75μg Vitamin D / 12mg tocopherol
  Arms: EPAVasc 2g; EPAVasc 2g x 2
Dietary Supplement: Corn Oil — Corn Oil
  Arms: Corn Oil

SUMMARY:
Investigation of the efficacy and safety of an Eicosapentaenoic acid (EPA) supplement versus a placebo supplement on plasma triglyceride levels as well as inflammatory, thrombotic, endothelial and platelet activation markers, in patients with type-2 diabetes mellitus (DM-2).

DETAILED DESCRIPTION:
The conflicting results of previous clinical trials regarding the clinical efficacy of omega-3 fatty acids, such as the STRENGTH and REDUCE-IT studies, as well as the published comments for the placebo used in the REDUCE-IT study (mineral oil), highlight the need for additional studies (pharmacodynamic, clinical, and basic research studies). The SEASIDE (Study of the Effect of Eicosapentaenoic acid, EPA, on Markers of Atherothrombosis in Patients with Type-2 Diabetes) is a phase 4 clinical study, aiming to investigate the efficacy of the dietary supplement EPAVasc, consisted of 1,875mg EPA / 125mg Docosahexaenoic acid (DHA) / 3.75μg Vitamin D / 12mg tocopherol, in reducing the plasma levels of triglycerides, markers of inflammation, coagulation, and platelet as well as endothelial functionality, in high or very high cardiovascular risk DM-2 patients, as compared with the administration of a placebo dietary supplement (Corn Oil). The safety of administering the above EPA supplementation to these patients will be also investigated. This study is expected to significantly advance the existing knowledge regarding the efficacy of EPA in reducing important cardiovascular risk biomarkers in high or very high cardiovascular risk DM-2 patients.

ELIGIBILITY:
Inclusion Criteria: The study will enroll DM-2 patients at high or very high cardiovascular risk, aged ≥ 50 years. Patients should have at least one additional cardiovascular risk factor (such as smoking, hypertension, HDL-cholesterol ≤40 mg/dL for Men, or ≤50mg/dL for Women, high-sensitivity C-reactive protein (hs-CRP)> 3mg/L, renal dysfunction (CrCl 30-60 mL/min), Ankle-Brachial Index (ABI) <0.9 (without symptoms of intermittent claudication). In addition, patients enrolled in the study will exhibit triglyceride levels >135 mg/dL and <500 mg/dL, despite adherence to the dietary recommendations given for their disease. These recommendations should be followed by all patients during the study. In addition to antidiabetic treatment, patients will receive statin or statin-ezetimibe combination therapy for at least 4 weeks prior to the first visit and should have LDL-cholesterol levels <100mg/dL. Antidiabetic and hypolipidemic treatment will remain unchanged during the study. All patients will sign a written informed consent prior to their inclusion in the study.

Exclusion Criteria

1. Patients with a history (≤ 12 months) of acute coronary syndrome (ACS) or ischemic stroke who are receiving antiplatelet therapy.
2. Patients with peripheral arterial disease or carotid artery disease (>50% stenosis by DOPPLER ultrasound criteria) receiving antiplatelet therapy.
3. Patients receiving monotherapy with any antiplatelet agent.
4. Patients with atrial fibrillation receiving any anticoagulation, or patients with a history of cardioembolic ischemic stroke or hemorrhagic stroke.
5. Patients with severe heart failure, (NYHA IV).
6. Patients with laboratory or clinically diagnosed severe active liver disease or liver failure (child-Pugh staging, score ≥ 5) or renal failure (eGFR < 30ml/min).
7. Patients with cancer, receiving any anticancer treatment.
8. Patients who are planned to undergo any surgical procedure.
9. Exclusion criteria will also include a. HbA1c levels >10.0%, b. history of acute or chronic pancreatitis, c. known hypersensitivity to fish or shellfish or to the components of the study product or placebo.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The percentage (%) change in plasma levels of triglycerides and markers of inflammation, coagulation, endothelial cell and platelet activation. | 3 months
  The primary composite efficacy endpoint is the percentage (%) change in each participant in plasma levels of triglycerides and markers of inflammation, coagulation, endothelial cell and platelet activation, comparing the placebo supplement and the investigating supplement.
Number of participants who suffer from bleeding events as defined by the Bleeding Academic Research Consortium (BARC) criteria during the entire follow-up period. | 3 months
  The Primary safety endpoint is major bleeding according to BARC (Bleeding Academic Research Consortium) criteria.

SECONDARY OUTCOMES:
The percentage (%) change in plasma levels of triglycerides. | 3 months
  The secondary efficacy endpoint is the (%) change in triglyceride levels of each participant.
The percentage (%) change in markers of inflammation. | 3 months
  The secondary efficacy endpoint is the (%) change in markers of inflammation, specifically Interleukin-1beta (IL-1β) (pg/ml) and Interleukin-6 (IL-6) (pg/ml).
The percentage (%) change in markers of coagulation. | 3 months
  The secondary efficacy endpoint is the (%) change in markers of coagulation specifically Tissue Factor (pg/ml) and Thrombin Time (sec).
The percentage (%) change in markers of endothelial cell activation. | 3 months
  The secondary efficacy endpoint is the (%) change in markers of endothelial cell activation specifically Monocyte Chemotactic Protein-1 (MCP-1) (pg/ml), Vascular Endothelial Cell Adhesion Molecule-1 (VCAM-1) (ng/mL) and von Willebrand Factor (vWF) (mIU/ml).
The percentage (%) change in markers of platelet activation. | 3 months
  The secondary efficacy endpoint is the (%) change in markers of platelet activation specifically soluble P-selectin (sP-selectin) (ng/ml), sCD40L (pg/ml) and Thromboxane A2 (TxA2) (pg/ml).
Number of participants who suffer from the secondary safety end points which are Atrial fibrillation, Palpitations, Arrhythmias, Heart failure, Pneumonia, Peripheral edema, Diarrhea. | 3 months
  Secondary safety endpoints are Atrial fibrillation, Palpitations, Arrhythmias, Heart failure, Pneumonia, Peripheral edema, Diarrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Atherothrombosis Research Centre / Laboratory of Biochemistry, University of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goel A, Pothineni NV, Singhal M, Paydak H, Saldeen T, Mehta JL. Fish, Fish Oils and Cardioprotection: Promise or Fish Tale? Int J Mol Sci. 2018 Nov 22;19(12):3703. doi: 10.3390/ijms19123703. PMID 30469489
- [Background] Innes JK, Calder PC. Marine Omega-3 (N-3) Fatty Acids for Cardiovascular Health: An Update for 2020. Int J Mol Sci. 2020 Feb 18;21(4):1362. doi: 10.3390/ijms21041362. PMID 32085487
- [Background] Cholewski M, Tomczykowa M, Tomczyk M. A Comprehensive Review of Chemistry, Sources and Bioavailability of Omega-3 Fatty Acids. Nutrients. 2018 Nov 4;10(11):1662. doi: 10.3390/nu10111662. PMID 30400360
- [Background] Yagi S, Fukuda D, Aihara KI, Akaike M, Shimabukuro M, Sata M. n-3 Polyunsaturated Fatty Acids: Promising Nutrients for Preventing Cardiovascular Disease. J Atheroscler Thromb. 2017 Oct 1;24(10):999-1010. doi: 10.5551/jat.RV17013. Epub 2017 Aug 24. PMID 28835582
- [Background] Maki KC, Johns C, Harris WS, Puder M, Freedman SD, Thorsteinsson T, Daak A, Rabinowicz AL, Sancilio FD. Bioequivalence Demonstration for Omega-3 Acid Ethyl Ester Formulations: Rationale for Modification of Current Guidance. Clin Ther. 2017 Mar;39(3):652-658. doi: 10.1016/j.clinthera.2017.01.019. Epub 2017 Feb 8. PMID 28189365
- [Background] de Carvalho CCCR, Caramujo MJ. The Various Roles of Fatty Acids. Molecules. 2018 Oct 9;23(10):2583. doi: 10.3390/molecules23102583. PMID 30304860
- [Background] Sherratt SCR, Juliano RA, Mason RP. Eicosapentaenoic acid (EPA) has optimal chain length and degree of unsaturation to inhibit oxidation of small dense LDL and membrane cholesterol domains as compared to related fatty acids in vitro. Biochim Biophys Acta Biomembr. 2020 Jul 1;1862(7):183254. doi: 10.1016/j.bbamem.2020.183254. Epub 2020 Mar 2. PMID 32135144
- [Background] Shibabaw T. Omega-3 polyunsaturated fatty acids: anti-inflammatory and anti-hypertriglyceridemia mechanisms in cardiovascular disease. Mol Cell Biochem. 2021 Feb;476(2):993-1003. doi: 10.1007/s11010-020-03965-7. Epub 2020 Nov 11. PMID 33179122
- [Background] Preston Mason R. New Insights into Mechanisms of Action for Omega-3 Fatty Acids in Atherothrombotic Cardiovascular Disease. Curr Atheroscler Rep. 2019 Jan 12;21(1):2. doi: 10.1007/s11883-019-0762-1. PMID 30637567
- [Background] Calder PC. Mechanisms of action of (n-3) fatty acids. J Nutr. 2012 Mar;142(3):592S-599S. doi: 10.3945/jn.111.155259. Epub 2012 Jan 25. PMID 22279140
- [Background] Kromhout D, Giltay EJ, Geleijnse JM; Alpha Omega Trial Group. n-3 fatty acids and cardiovascular events after myocardial infarction. N Engl J Med. 2010 Nov 18;363(21):2015-26. doi: 10.1056/NEJMoa1003603. Epub 2010 Aug 28. PMID 20929341
- [Background] ASCEND Study Collaborative Group; Bowman L, Mafham M, Wallendszus K, Stevens W, Buck G, Barton J, Murphy K, Aung T, Haynes R, Cox J, Murawska A, Young A, Lay M, Chen F, Sammons E, Waters E, Adler A, Bodansky J, Farmer A, McPherson R, Neil A, Simpson D, Peto R, Baigent C, Collins R, Parish S, Armitage J. Effects of n-3 Fatty Acid Supplements in Diabetes Mellitus. N Engl J Med. 2018 Oct 18;379(16):1540-1550. doi: 10.1056/NEJMoa1804989. Epub 2018 Aug 26. PMID 30146932
- [Background] Manson JE, Cook NR, Lee IM, Christen W, Bassuk SS, Mora S, Gibson H, Albert CM, Gordon D, Copeland T, D'Agostino D, Friedenberg G, Ridge C, Bubes V, Giovannucci EL, Willett WC, Buring JE; VITAL Research Group. Marine n-3 Fatty Acids and Prevention of Cardiovascular Disease and Cancer. N Engl J Med. 2019 Jan 3;380(1):23-32. doi: 10.1056/NEJMoa1811403. Epub 2018 Nov 10. PMID 30415637
- [Background] Fialkow J. Omega-3 Fatty Acid Formulations in Cardiovascular Disease: Dietary Supplements are Not Substitutes for Prescription Products. Am J Cardiovasc Drugs. 2016 Aug;16(4):229-239. doi: 10.1007/s40256-016-0170-7. PMID 27138439
- [Background] Nicholls SJ, Lincoff AM, Garcia M, Bash D, Ballantyne CM, Barter PJ, Davidson MH, Kastelein JJP, Koenig W, McGuire DK, Mozaffarian D, Ridker PM, Ray KK, Katona BG, Himmelmann A, Loss LE, Rensfeldt M, Lundstrom T, Agrawal R, Menon V, Wolski K, Nissen SE. Effect of High-Dose Omega-3 Fatty Acids vs Corn Oil on Major Adverse Cardiovascular Events in Patients at High Cardiovascular Risk: The STRENGTH Randomized Clinical Trial. JAMA. 2020 Dec 8;324(22):2268-2280. doi: 10.1001/jama.2020.22258. PMID 33190147
- [Background] Budoff MJ, Bhatt DL, Kinninger A, Lakshmanan S, Muhlestein JB, Le VT, May HT, Shaikh K, Shekar C, Roy SK, Tayek J, Nelson JR. Effect of icosapent ethyl on progression of coronary atherosclerosis in patients with elevated triglycerides on statin therapy: final results of the EVAPORATE trial. Eur Heart J. 2020 Oct 21;41(40):3925-3932. doi: 10.1093/eurheartj/ehaa652. PMID 32860032
- [Background] Watanabe T, Ando K, Daidoji H, Otaki Y, Sugawara S, Matsui M, Ikeno E, Hirono O, Miyawaki H, Yashiro Y, Nishiyama S, Arimoto T, Takahashi H, Shishido T, Miyashita T, Miyamoto T, Kubota I; CHERRY study investigators. A randomized controlled trial of eicosapentaenoic acid in patients with coronary heart disease on statins. J Cardiol. 2017 Dec;70(6):537-544. doi: 10.1016/j.jjcc.2017.07.007. Epub 2017 Aug 31. PMID 28863874
- [Background] Bhatt DL, Steg PG, Miller M, Brinton EA, Jacobson TA, Ketchum SB, Doyle RT Jr, Juliano RA, Jiao L, Granowitz C, Tardif JC, Ballantyne CM; REDUCE-IT Investigators. Cardiovascular Risk Reduction with Icosapent Ethyl for Hypertriglyceridemia. N Engl J Med. 2019 Jan 3;380(1):11-22. doi: 10.1056/NEJMoa1812792. Epub 2018 Nov 10. PMID 30415628
- [Background] Tsoumani ME, Kalantzi KI, Dimitriou AA, Ntalas IV, Goudevenos IA, Tselepis AD. Antiplatelet efficacy of long-term treatment with clopidogrel besylate in patients with a history of acute coronary syndrome: comparison with clopidogrel hydrogen sulfate. Angiology. 2012 Oct;63(7):547-51. doi: 10.1177/0003319711427697. Epub 2011 Dec 5. PMID 22144668
- [Background] Ntalas IV, Kalantzi KI, Tsoumani ME, Vakalis JN, Vasilakopoulos V, Vardakis K, Vemmos KN, Voukelatou M, Giannakoulas G, Giatrakos I, Giogiakas V, Goumas G, Dimoulis N, Draganigos A, Efthimiadis I, Thoma M, Kazakos E, Kipouridis N, Konstantinou S, Bourdakis A, Nikolopoulos D, Peltekis L, Prokopakis N, Sinteles I, Stroumbis CS, Terzoudi K, Tsilias K, Xaraktsis I, Charmpas C, Hatziathanasiou G, Christogiannis Z, Panagiotakos DB, Goudevenos JA, Tselepis AD. Generic Clopidogrel Besylate in the Secondary Prevention of Atherothrombotic Events: A 6-month Follow-up of a Randomised Clinical Trial. Curr Vasc Pharmacol. 2015;13(6):809-18. doi: 10.2174/1570161113666150316220515. PMID 25782408
- [Background] Ntalas IV, Kalantzi KI, Tsoumani ME, Bourdakis A, Charmpas C, Christogiannis Z, Dimoulis N, Draganigos A, Efthimiadis I, Giannakoulas G, Giatrakos I, Giogiakas V, Goumas G, Hatziathanasiou G, Kazakos E, Kipouridis N, Konstantinou S, Milionis H, Nikolopoulos D, Peltekis L, Prokopakis N, Sinteles I, Stroumbis C, Terzoudi K, Thoma M, Tsilias K, Vakalis I, Vardakis K, Vasilakopoulos V, Vemmos K, Voukelatou M, Xaraktsis I, Panagiotakos DB, Goudevenos JA, Tselepis AD. Salts of Clopidogrel: Investigation to Ensure Clinical Equivalence: A 12-Month Randomized Clinical Trial. J Cardiovasc Pharmacol Ther. 2016 Nov;21(6):516-525. doi: 10.1177/1074248416644343. Epub 2016 Apr 14. PMID 27081185
- [Background] Kalantzi K, Tentolouris N, Melidonis AJ, Papadaki S, Peroulis M, Amantos KA, Andreopoulos G, Bellos GI, Boutel D, Bristianou M, Chrisis D, Dimitsikoglou NA, Doupis J, Georgopoulou C, Gkintikas SA, Iraklianou S, Kanellas Kappa, Kotsa K, Koufakis T, Kouroglou M, Koutsovasilis AG, Lanaras L, Liouri E, Lixouriotis C, Lykoudi A, Mandalaki E, Papageorgiou E, Papanas N, Rigas S, Stamatelatou MI, Triantafyllidis I, Trikkalinou A, Tsouka AN, Zacharopoulou O, Zoupas C, Tsolakis I, Tselepis AD. Efficacy and Safety of Adjunctive Cilostazol to Clopidogrel-Treated Diabetic Patients With Symptomatic Lower Extremity Artery Disease in the Prevention of Ischemic Vascular Events. J Am Heart Assoc. 2021 Jan 5;10(1):e018184. doi: 10.1161/JAHA.120.018184. Epub 2020 Dec 17. PMID 33327737
- [Background] Tsoumani ME, Kalantzi KI, Dimitriou AA, Ntalas IV, Goudevenos IA, Tselepis AD. Effect of clopidogrel besylate on platelet reactivity in patients with acute coronary syndromes. Comparison with clopidogrel hydrogen sulfate. Expert Opin Pharmacother. 2012 Feb;13(2):149-58. doi: 10.1517/14656566.2012.644536. Epub 2011 Dec 21. PMID 22188544
- [Background] Woodman RJ, Mori TA, Burke V, Puddey IB, Watts GF, Beilin LJ. Effects of purified eicosapentaenoic and docosahexaenoic acids on glycemic control, blood pressure, and serum lipids in type 2 diabetic patients with treated hypertension. Am J Clin Nutr. 2002 Nov;76(5):1007-15. doi: 10.1093/ajcn/76.5.1007. PMID 12399272
- [Background] Ryan, Thomas P. 2013. Sample Size Determination and Power. John Wiley & Sons. New Jersey.
- [Background] Harden M, Friede T. Sample size calculation in multi-centre clinical trials. BMC Med Res Methodol. 2018 Nov 29;18(1):156. doi: 10.1186/s12874-018-0602-y. PMID 30497390
- [Background] Liu Y, Xu H. Sample size re-estimation for pivotal clinical trials. Contemp Clin Trials. 2021 Mar;102:106215. doi: 10.1016/j.cct.2020.106215. Epub 2020 Nov 18. PMID 33217555
- [Background] Wang P, Chow SC. Sample size re-estimation in clinical trials. Stat Med. 2021 Nov 30;40(27):6133-6149. doi: 10.1002/sim.9175. Epub 2021 Aug 25. PMID 34433225
- [Background] Grayling MJ, Mander AP, Wason JMS. Blinded and unblinded sample size reestimation in crossover trials balanced for period. Biom J. 2018 Sep;60(5):917-933. doi: 10.1002/bimj.201700092. Epub 2018 Aug 3. PMID 30073679
- [Background] Yokoyama M, Origasa H, Matsuzaki M, Matsuzawa Y, Saito Y, Ishikawa Y, Oikawa S, Sasaki J, Hishida H, Itakura H, Kita T, Kitabatake A, Nakaya N, Sakata T, Shimada K, Shirato K; Japan EPA lipid intervention study (JELIS) Investigators. Effects of eicosapentaenoic acid on major coronary events in hypercholesterolaemic patients (JELIS): a randomised open-label, blinded endpoint analysis. Lancet. 2007 Mar 31;369(9567):1090-8. doi: 10.1016/S0140-6736(07)60527-3. PMID 17398308